CLINICAL TRIAL: NCT02287194
Title: Clinical Registry of Cholangioscopy Using the SpyGlass™ Direct Visualization System Throughout China
Brief Title: SpyGlass Direct Visualization System Clinical Registry in China
Acronym: SpyChina
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: E7101
Record Dates: First submitted 2014-08-20; First posted 2014-11-10 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2017-09

CONDITIONS: Biliary Tract Diseases
MeSH Terms: conditions — Biliary Tract Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SpyGlass Direct Visualization System: Any patient who has undergone SpyGlass Choledochoscopy procedures for diagnosis and/or treatment of biliary tract diseases.
  Interventions: Device: SpyGlass

INTERVENTIONS:
Device: SpyGlass — The SpyGlass Direct Visualization System is an integrated product platform that is designed to provide a direct intraluminal view of the biliary duct system and direct therapeutic devices.

SUMMARY:
To document indications for cholangioscopy and clinical utility of the SpyGlass Direct Visualization System in China when used per standard of practice.

Prospective, Post market, Multi-center, Non-randomized Study

DETAILED DESCRIPTION:
Patients who presenting with an indication for cholangioscopy or presenting with a possible indication for cholangioscopy to be determined during the ERCP procedure immediately preceding the SpyGlass procedure will join this study, totally 500 patients across 16 sites throughout China will participate in study. After SpyGlass operation, all patients will be followed for 72 hours to observe adverse events, and patients with indeterminate stricture or undefined filling defect indication with tissue sampling not yielding histopathology positive for malignancy and unresolved device and/or procedure related SAE at 72 Hours will continue to be followed up until 6 months. Finally, procedure success rate will be analyzed as primary endpoint, and SAEs and impact of patients management will be analyzed as secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 and not above 85.
2. Willing and able to provide written informed consent to participate in the study.
3. Willing and able to comply with the study procedures.
4. Indicated for ERCP and cholangioscopy or indicated for ERCP with suspected need for cholangioscopy.

Exclusion Criteria:

1. Endoscopic techniques are contraindicated.
2. ERCP is contraindicated
3. A medical condition that warrants the use of the device outside of the indication for use.
4. Requirement for anticoagulation that cannot be safely stopped at least 7 days prior to the procedure.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients seen at an investigational site during the enrollment period
  * Presenting with an indication for cholangioscopy, or
  * Presenting with a possible indication for cholangioscopy to be determined during the ERCP procedure immediately preceding the SpyGlass procedure.
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2014-11-28 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Procedural success rate | 72 hours
  1. For indeterminate strictures or undefined filling defects cases procedural success is defined as 1) ability to visualize stricture or defect, and 2) ability to provide visual impression of malignancy, and 3) when applicable, ability to obtain SpyBite biopsy adequate for histology
  2. For biliary stone cases procedural success is defined as 1) ability to visualize the stone(s), and 2) ability to successfully initiate stone fragmentation, and 3) ability to achieve stone clearance in one or more SpyGlass procedures.
  3. For other indications procedural success is defined as ability to establish diagnosis and /or complete therapy in the following categories: 1) pre-operative assessment of extent of peri-ampullary and biliary tumors, 2) selective guidewire placement, 3) assessment of unexplained hemobilia, 4) assessment of portal biliopathy, 5) assessment of intraductal biliary ablation therapy, 6) extraction of migrated stents, or 7) other.

SECONDARY OUTCOMES:
Safety Endpoints | Post Procedure
  Evaluation of serious adverse events (SAEs) related to the SpyGlass devices and/or the SpyGlass procedure from enrollment through the 72 Hour Post Procedure Follow-up Visit.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, Prof., Principal Investigator — Changhai Hospital
Locations (1):
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen YK. Preclinical characterization of the Spyglass peroral cholangiopancreatoscopy system for direct access, visualization, and biopsy. Gastrointest Endosc. 2007 Feb;65(2):303-11. doi: 10.1016/j.gie.2006.07.048. PMID 17258991